CLINICAL TRIAL: NCT07011186
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of TQB3909 Tablets in Combination With Azacitidine in Subjects With Myeloid Malignancies
Brief Title: A Clinical Trial of TQB3909 Tablets in Combination With Azacitidine for the Treatment of Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-Ib/II-03
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-03

CONDITIONS: Myeloid Malignancy
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3909 Tablets + Azacitidine (Experimental): TQB3909 Tablets administered once-daily. 28 days as a treatment cycle.
  Interventions: Drug: TQB3909 Tablets + Azacitidine

INTERVENTIONS:
Drug: TQB3909 Tablets + Azacitidine — TQB3909 is a protein inhibitor; Azacitidine is a cytidine nucleoside analogue

SUMMARY:
This is an open, multi-center clinical study designed to evaluate the safety, tolerability and efficacy of TQB3909 tablets in combination with azacitidine in subjects with myeloid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and signed informed consent, good compliance
* Age: ≥18 years old (at the time of signing the informed consent); expected survival time greater than 3 months.
* Diagnosis of one of the following diseases:

  1. Acute Myeloid Leukemia (AML):
  2. Myelodysplastic Syndromes (MDS)
  3. Major organ functions are normal.
  4. Fertile male and female subjects agree to use contraception during the study and for 6 months after the study ends.

Exclusion Criteria:

* Comorbidities and Medical History:

  1. Diagnosis of or current concomitant malignancy within 3 years prior to the first dose;
  2. Presence of multiple factors affecting oral drug intake and/or absorption;
  3. Major surgical procedures or significant traumatic injuries within 28 days prior to the first dose;
  4. History of arterial/venous thrombotic events within 6 months prior to the first dose;
  5. History of psychiatric drug abuse that cannot be discontinued, or psychiatric disorders;
  6. Presence of any severe and/or uncontrolled disease in the subject.
* Tumor-related Symptoms and Treatment:

  1. Diagnosis of Acute Promyelocytic Leukemia (APL), Myelodysplastic Syndromes/Myeloproliferative Neoplasms (MDS/MPN);
  2. Presence of leukemia central nervous system (CNS) involvement or high suspicion of CNS involvement but unable to confirm;
  3. Subjects with extramedullary disease only in AML;
  4. Presence of life-threatening severe leukemia-related complications;
* Study Treatment-related:

  1. Received live vaccines within 4 weeks prior to the first dose, or planned to receive live vaccines during the study period;
  2. Participated in other clinical trials involving anti-tumor drugs within 4 weeks prior to the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) and serious adverse events (SAE), abnormal laboratory parameters | Up to 24 weeks
  Any adverse medical event that occurred from the time the subject signed the informed consent until 28 days after the last dose/start of the new antitumor therapy (whichever occurs first)
Complete Remission + Complete Remission with Partial Hematologic Recovery (CR+CRh) Rate | Up to 4 weeks
  Complete Remission + Complete Remission with Partial Hematologic Recovery (CR+CRh) Rate

SECONDARY OUTCOMES:
Acute Myeloid Leukemia: Investigator-Assessed Objective Response Rate (ORR) | Up to 4 weeks
  Proportion of subjects with best response as Complete Remission (CR), Complete Remission with Incomplete Hematologic Recovery (CRi), Morphologic Leukemia-Free State (MLFS), or Partial Remission (PR)
Myelodysplastic Syndromes: Investigator-Assessed Objective Response Rate (ORR) | Up to 4 weeks
  Proportion of subjects with best response as CR, Morphological Complete Remission (mCR), or PR
Acute Myeloid Leukemia: Complete Remission + Complete Remission with Incomplete Hematologic Recovery (CR+CRi) Rate | Up to 4 weeks
  Proportion of subjects with best response as CR+CRi. CRi refers to meeting all CR criteria except for residual neutrophil count decrease (ANC < 1.0 × 109/L) or platelet count decrease (PLT < 100 × 109/L).
Acute Myeloid Leukemia: Complete Remission + Complete Remission with Partial Hematologic Recovery (CR+CRh) Rate | Up to 4 weeks
  Proportion of subjects with best response as CR
Acute Myeloid Leukemia and Myelodysplastic Syndromes: Complete Remission (CR) Rate | Up to 4 weeks
  Proportion of subjects with best response as CR
Acute Myeloid Leukemia: Duration of Remission (DOR) | Up to 4 weeks
  For all subjects with best response as CR, CRi, MLFS, or PR, the time from the first date of achieving remission to the first recorded date of disease progression, relapse, or death (whichever occurs first).
Acute Myeloid Leukemia: Duration of CR + CRh (DOCR+CRh) | Up to 4 weeks
  For all subjects with best response as CR or CRh, the time from the first date of achieving CR or CRh to the first recorded date of relapse or death (whichever occurs first).
Acute Myeloid Leukemia: Duration of Complete Remission (DOCR) | Up to 4 weeks
  For all subjects with best response as CR, the time from the first date of achieving CR to the first recorded date of relapse or death (whichever occurs first).
Acute Myeloid Leukemia: Time to First Complete Remission (TTCR) | Up to 4 weeks
  For all subjects with best response as CR or CRh, the time from the first date of medication to the first date of CR or CRh.
Acute Myeloid Leukemia: Time to First Complete Remission (TTCR) | Up to 4 weeks
  For subjects with best response as CR, the time from the first date of medication to the first date of CR.
Acute Myeloid Leukemia and Myelodysplastic Syndromes: Event-Free Survival (EFS) | Up to 4 weeks
  Defined as the duration from the first dose of medication to treatment failure, relapse after CR or CRi, or death due to any cause (whichever occurs first). Treatment failure is defined as not achieving CR or CRi at any assessment time during treatment. Subjects with treatment failure will be considered to have an EFS event on the first day after the first dose. For subjects with CR or CRi, the event time will be the time of disease relapse or death (whichever occurs first).
Acute Myeloid Leukemia and Myelodysplastic Syndromes: Overall Survival (OS) | Up to 60 weeks
  The time from the first dose of medication to the date of death due to any cause.
Myelodysplastic Syndromes: Hematologic Improvement (HI) Rate | Up to 4 weeks
  Proportion of subjects meeting Hematologic Improvement (HI) criteria, including Hematologic Improvement - Erythrocyte (HI-E), Hematologic Improvement - Platelet (HI-P), and Hematologic Improvement - Neutrophil (HI-N).
Myelodysplastic Syndromes: Transfusion Independence Rate | Up to 8 weeks
  The proportion of subjects who did not require transfusions for at least 56 days after baseline, relative to the number of baseline transfusion-dependent and transfusion-independent subjects.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Beijing Chaoyang Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Harbin The First Hospital, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Zhuzhou Central Hospita, Zhuzhou, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Tai'an Central Hospital (Tai'an Central Hospital affiliated to Qingdao University, Mount Taishan Medical Center), Taian, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - ShangHai Tongren Hospital, Shanghai, Shanghai Municipality
  - Shanghai Yueyang Integrated Traditional Chinese Medicine and Western Medicine Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality
  - People's hospital of deyang city, Deyang, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - People's Hospital of Tianjin (City), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang